CLINICAL TRIAL: NCT06714695
Title: Evaluation of the Effective Concentration of Chitosan Mouthwash on the Recurrence of Black Stains in Pediatric Patients. a Crossover Controlled Clinical Trial
Brief Title: A Crossover Clinical Study to Evaluate the Effect of Chitosan Mouthwash on Recurrence of Black Stains in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Rawda wagih Mostafa Hassan, Doctorate candidate in faculty of dental medicine Azhar university girls, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: (P-PE-22-03)
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Black Stains
Keywords: Black stains; chromogenic; Children; Pediatric; Recurrence
MeSH Terms: conditions — Recurrence | interventions — Chitosan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pediatric patients before and after using chitosan mouthwash (Other): pediatric patients with black stains will be recruited in the study. Scaling and polishing will be done then followed up for 3 months, then scaling and polishing will be repeated after follow up period and the patient will be given chitosan mouthwash to be used for additional 3 months.
  Interventions: Drug: Chitosan

INTERVENTIONS:
Drug: Chitosan — chitosan mouthwash

SUMMARY:
The goal of this clinical trial is to learn if Chitosan mouthwash works to affect the recurrence of black stains in pediatric patients. The main questions it aims to answer are:

Does Chitosan mouthwash lower the number of times participants need to do a scaling and polishing cleaning sessions more than normal? Does Chitosan mouthwash will decrease the recurrence of black stains in children and improve esthetics ?

Participants will:

Take chitosan every day for 4 months Visit the clinic once every 6 weeks for checkups and data collection

ELIGIBILITY:
Inclusion Criteria:

* 1. Cooperative child to be able to perform and tolerate different oral hygiene procedures 2. Parents providing informed consent 3. Accept 18 weeks follow up period 4. Teeth showing black stains without calculus.

Exclusion Criteria:

* 1. Patients with Allergic reactions to food & drugs containing derivatives from crustacean organisms. 2. Taking any antibiotic drugs within 2- week period before sample collection. 3. Taking any dietary supplements containing iron. 4. Teeth selected should be free of caries 5. Free of any developmental defects

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Black stains | 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dental medicine Azhar University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Milleman KR, Creeth JE, Burnett GR, Milleman JL. A randomized clinical trial to evaluate the stain removal efficacy of a sodium phytate dentifrice formulation. J Esthet Restor Dent. 2018 Mar;30(2):E45-E51. doi: 10.1111/jerd.12355. Epub 2018 Feb 7. PMID 29411532
- [Background] Qin C, Li H., Xiao Q, Liu Y, Zhu J, Du Y. Water-solubility of chitosan and its antimicrobial activity, Carbohydr Polyr 2006; 63:367-74.
- [Background] Koch MJ, Bove M, Schroff J, Perlea P, Garcia-Godoy F, Staehle HJ. Black stain and dental caries in schoolchildren in Potenza, Italy. ASDC J Dent Child. 2001 Sep-Dec;68(5-6):353-5, 302. PMID 11985199